CLINICAL TRIAL: NCT01175304
Title: Study of Sleep Habits and Prevalence of Sleepiness in a Health Care Environment in Barcelona
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Patricia Lloberes MD, phD, Servei Pneumologia Vall d'Hebron
Other Study IDs: PR(AG)40/2009
Record Dates: First submitted 2010-07-27; First posted 2010-08-04 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-07

CONDITIONS: Sleep; Subjective Sleepiness; Sleep Apnea
Keywords: sleep; sleep apnea; work; sleep habits; sleepiness
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleepiness

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Workers in a Barcelona tertiary hospital: Workers attending annual medical checkups

SUMMARY:
The purpose of this study is the description of sleeping habits in a working population in the investigators health care environment, analyzing the prevalence of daytime sleepiness and symptoms compatible with the sleep apnea syndrome and finally to analyze predictors of daytime sleepiness.

DETAILED DESCRIPTION:
Descriptive study population in a working population in a tertiary hospital in Barcelona (Spain). The population will consist of subjects who come to the annual medical checkups at the hospital. Exclusion criteria: pregnant women.

Assuming a prevalence of excessive daytime sleepiness of 20 ± 5% with a confidence interval of 95% the number of subjects to be studied is 500.

Methods:

1. General information and anthropometric data
2. Questionnaires

2.1. General questionnaire, working schedules and anthropometric data

2.2. Sleeping habits questionnaire

2.3. Frequency of perceived daytime sleepiness (5 item questionnaire(Kim H, Young T.Sleep 2005;28:625-634)

1. Not rested during the day no matter how many hours of sleep you had
2. Feeling of excessive daytime sleepiness 0.71† 0.08 0.03
3. Great difficulty getting up in the morning 0.62† -0.06 -0.05
4. Need for coffee, or other stimulants to stay awake during the day
5. Falling asleep or dozing momentarily at meetings, church, etc. (item responses (frequency per month): 0=never, 1=rarely (once), 2= sometimes(2-4), 3 (often (5-15), 4=almost always (16-30)

2.4. Epworth sleepiness scale

2.5. Berlin Questionnaire

Questionnaires will be answered in an anonymous and voluntary way on the part of workers.

Data analysis:

1. General and anthropometric data (Mean and Standard Deviation)
2. Sleep habits: sleep latency, sleep time (night and 24 hours), satisfaction with sleep, sleep-debt, anxiolytic medication before bedtime
3. Prevalence of daytime sleepiness:

   * Daytime sleepiness questionnaire, consisting of five items coded on a 0-4 ordinal scale (range 00-20 final score).
   * Epworth sleepiness scale: range 0-24, being a value ≥ 10 indicative of daytime sleepiness.
   * Association between daytime sleepiness, anthropometric variables, and variables derived from sleeping habits questionnaire.
4. Prevalence of traffic accidents in itinera, and their association with daytime sleepiness, shift work or sleep apnea symptoms.
5. Berlin Questionnaire: - Category 1 positive with 2 or more positive answers to questions 2-6 - Category 2 positive with 2 or more positive answers to questions 7-9 - Category 3 positive response with a positive and / or a BMI> 30 or more positive categories indicates a high probability of sleep apnea syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Workers attending annual checkups at the Hospital's medical department.

Exclusion Criteria:

* Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample of 500 consecutive tertiary hospital workers in the city of Barcelona (Spain), attending annual checkups at the Hospital's medical department.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2010-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Sleeping time and sleeping schedules in a working population in a health care environment | 4 months
  Number of hours of sleep during the working days and during the weekend

SECONDARY OUTCOMES:
Symptoms compatible with the sleep apnea syndrome | 4 months
  Results of the Berlin Questionnaire
Analyze predictors of daytime sleepiness | 4 months
  Anhropometric, hours of sleep and Berlin questionnaires variables
Frequency of perceived daytime sleepiness | 4 months
  Scores of sleepiness questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Lloberes, MD,pHD, Principal Investigator — Servei de Pneumologia Hospital Universitari Vall d'Hebron Barcelona
Locations (1):
- Hospital Universitari Vall D' Hebron, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Kaneita Y, Ohida T, Uchiyama M, Takemura S, Kawahara K, Yokoyama E, Miyake T, Harano S, Suzuki K, Yagi Y, Kaneko A, Tsutsui T, Akashiba T. Excessive daytime sleepiness among the Japanese general population. J Epidemiol. 2005 Jan;15(1):1-8. doi: 10.2188/jea.15.1. PMID 15678919
- [Background] Kim H, Young T. Subjective daytime sleepiness: dimensions and correlates in the general population. Sleep. 2005 May;28(5):625-34. doi: 10.1093/sleep/28.5.625. PMID 16171277
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Netzer NC, Hoegel JJ, Loube D, Netzer CM, Hay B, Alvarez-Sala R, Strohl KP; Sleep in Primary Care International Study Group. Prevalence of symptoms and risk of sleep apnea in primary care. Chest. 2003 Oct;124(4):1406-14. doi: 10.1378/chest.124.4.1406. PMID 14555573